CLINICAL TRIAL: NCT01980758
Title: Pilot Study of Laparoscopic Gastric Plication in Adolescents With Severe Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Children's Hospital of Richmond (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM14809
Record Dates: First submitted 2013-09-26; First posted 2013-11-11 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Obesity
Keywords: obesity, pediatric obesity, bariatric, bariatric surgery
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery (Experimental): Laparoscopic Gastric Plication
  Interventions: Procedure: Laparoscopic Gastric Plication

INTERVENTIONS:
Procedure: Laparoscopic Gastric Plication — The study will examine the effects of a type of weight loss surgery on obese adolescents age 14-19. ) The study protocol includes pre-treatment assessments followed by a 2-month education and lifestyle modification treatment program. Following surgery, comprehensive follow-up care will be provided over a 3 year period.

SUMMARY:
The proposed study aims to investigate the effects of laparoscopic gastric plication (LGP) on excess body weight, body mass index, and weight-related medical and psychological co-morbidities in obese adolescents. Additionally, we will evaluate the safety and efficacy of this procedure (implemented within a multidisciplinary comprehensive lifestyle modification program) on changes in the patients' medical status, psychosocial and psychological functioning, physical fitness, and health-related quality of life.

Study hypothesis:

1. Laparoscopic gastric plication performed on carefully selected obese adolescents within a multidisciplinary treatment program providing pre and post-surgical behavioral and psychological support and education will result in: a) initial and sustained reductions in excess body weight and body mass index, b) improvements in psychological functioning, physical fitness, and health-related quality of life, and c) reduction in weight-related comorbidities.
2. LGP will be a safe procedure, with complication rates that are comparable to or lower than what has been found in other published reports of surgical weight loss procedures used in obese adolescents.

DETAILED DESCRIPTION:
The complete study protocol, which is described in detail below, spans 3 years and includes 11 research assessment points (Pre-1, Pre-2, T0, T1, T2, T3, T4, T5, T6, T7, and T8). Please refer to Figure 2. Study Protocol from Enrollment to Post-Surgical Assessments. Select pre-treatment assessments will be conducted initially (Pre-1), followed by a 2-month pre-surgical education and lifestyle modification treatment program, consisting of four visits with psychology, nutrition, exercise, and surgery. After successful completion of this pre-surgical education program, a more comprehensive pre-surgical assessment by a surgeon (Pre-2) will be conducted. If patients decide to pursue the study, in the two weeks prior to surgery, participants will be asked to adhere to a pre-surgical diet, exclusion and inclusion criteria will be reviewed again by the study team, and verbal consent/assent will be re-confirmed with adolescents and parent(s). Following surgery (T0), comprehensive follow-up care will be provided via the multidisciplinary team at the Healthy Lifestyles Center (HLC) at Children's Hospital of Richmond at Virginia Commonwealth University (CHoR at VCU). The follow-up period will be divided into three phases: 1) Early Post-Operative Phase (0-5 months), 2) Late Post-Operative phase (6-12 months), and 3) Long-term Follow-up Phase (13-36 months). In conjunction with clinical follow-up, repeat standardized research assessments will be conducted post-operatively at 1-2 weeks (T1), 6 weeks (T2), 3 months (T3), 6 months (T4), 12 months (T5), 18 months (T6), 24 months (T7), and 36 months (T8). Specific screening, pre-surgical, perioperative, and post-surgical study procedures at each time point are described fully below and outlined in Figure 2 and Table 1. Additionally, all research measures are described in detail in the Measures Section. If any participant requires any additional visit during the time of this study, data from these visits will also be collected for this study. Care directly related to the surgery and study will not be billed but other medical issues such as hypertension, diabetes, hypercholesterolemia and depression may require management outside of the scope of the study and will be billed accordingly

ELIGIBILITY:
Inclusion Criteria:

* Age 14 - 19.
* At physical maturity.
* BMI of greater than or equal to 35 kg/m2 with major comorbidities, or BMI of greater than 40 kg/m2 with other weight related comorbidities.
* Must have undergone comprehensive pre-surgical assessments by a multi-disciplinary team.
* Must have at least 6 months of medically observed and attempted non-surgical weight loss.
* Must have demonstrated suboptimal weight loss following participation in a lifestyle intervention.
* Must have parents involved in all phases of recruitment and intervention.

Exclusion Criteria:

* Underlying genetic or endocrine disorder, which would preclude weight loss through behavioral and surgical techniques.
* Less than six months of participation in a medically-supervised weight management efforts.
* Active untreated, unstable psychopathology (to include active psychosis, severe depression, or significant eating pathology), as determined by psychological evaluation.
* Active suicidal ideation, as determined by psychological evaluation.
* Inadequate social support, as determined by psychological evaluation.
* Inability to provide informed consent/assent, as evidenced by clinical interview and cognitive assessments.
* Severe mental retardation, as evidenced by clinical interview and cognitive assessments.
* Demonstrated pattern of poor adherence to medical regimen and lifestyle modification.
* Active substance abuse, including tobacco use, as demonstrated by clinical interview and psychological evaluation. Inadequate knowledge of risks and patient responsibilities, as determined by clinical interview and knowledge quiz.
* Reported pregnancy within the past year, current pregnancy, or planning to become pregnant in the next three years.
* History or clinical symptoms of severe gastrointestinal reflux disease (GERD)
* Person is not deemed for medical reasons to be a surgical candidate.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Reduction of Excess Body Weight | 6 months post-surgery

SECONDARY OUTCOMES:
Reduction in comorbidities to obesity | 6 months
Changes in lifestyle choices | 1 year
Improvement in quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Lanning, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU, Richmond, Virginia, United States